CLINICAL TRIAL: NCT00603499
Title: Hypomagnesemia as a Risk Factor for Development of Metabolic Syndrome
Brief Title: Magnesium and Metabolic Syndrome
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Instituto Mexicano del Seguro Social (Other Government)
Responsible Party: Fernando Guerrero-Romero, Biomedical Research Unit, Instituto Mexicano del Seguro Social
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2000-161-0027; IMSS
Record Dates: First submitted 2008-01-16; First posted 2008-01-29 (Estimated); Last update posted 2008-01-29 (Estimated); Status verified 2008-01

CONDITIONS: Diabetes Mellitus; High Blood Pressure; Hypomagnesemia
Keywords: Diabetes; Hypertension; Hypomagnesemia
MeSH Terms: conditions — Diabetes Mellitus; Hypertension | interventions — Magnesium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Magnesium chloride
  Interventions: Dietary Supplement: Magnesium chloride
- 2 (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Magnesium chloride — Subjects in the intervention group received 2.5 gr of MgCl2 daily during 4 months, from a solution solution containing 50 gr of MgCl2 by 1000 ml.
  Arms: 1
Other: Placebo — Subjects in the control group received inert placebo once per day during 4 months
  Arms: 2

SUMMARY:
Objective : to test the BP lowering-effect of oral magnesium supplementation, as magnesium chloride (MgCl2) solution, 2.5 g daily, in uncomplicated hypertensive type 2 diabetic subjects with decreased serum magnesium levels Design : Randomised double blind placebo controlled trial. Setting : Outpatients with type 2 diabetes from Durango, city in northern Mexico Subjects : 82 subjects between 40 and 75 years of age with type 2 diabetes serum magnesium deficiency and uncomplicated hypertension.

Interventions : During 4 months the intervention group received 2.5 gr of magnesium chloride (50 ml of a solution containing 50 gr of MgCl2 by 1000 ml of solution ). Controls received inert placebo.

Main outcome measure: Change in blood pressure. Increase of serum magnesium Secondary outcomes measures: Changes in lipid profile

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* Decreased serum magnesium levels
* Uncomplicated hypertension
* 40 and 75 years of age
* Men and Women

Exclusion Criteria:

* Chronic diarrhea
* Alcohol intake (equal or more than 30 g per day)
* Use of diuretics and/or calcium antagonists drugs
* Previous oral magnesium supplementation
* Ischemic diseases; AND
* Reduced renal function

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2006-07; Primary Completion 2007-08 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Reduction in the systolic and diastolic blood pressures | 2 y

SECONDARY OUTCOMES:
Average increase of serum magnesium levels Changes in lipid profile | 2 y

CONTACTS AND LOCATIONS:
Overall Officials: Martha Rodriguez-Moran, MD, MSc, PhD, Principal Investigator — Instituto Mexicano del Seguro Social
Locations (1):
- Biomedical Research Unit, Durango, Durango, Mexico